CLINICAL TRIAL: NCT02675270
Title: Rehabilitation and Prophylaxis of Anomia in Primary Progressive Aphasia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Georgetown University (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH); National Institute on Aging (NIA) (NIH); Johns Hopkins University (Other)
Responsible Party: Principal Investigator, Aaron Meyer, PhD, Assistant Professor, Georgetown University
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: R01DC011317 (NIH)
Record Dates: First submitted 2016-01-28; First posted 2016-02-05 (Estimated); Last update posted 2024-09-25 (Actual); Status verified 2024-09

CONDITIONS: Aphasia, Primary Progressive; Anomia; Alzheimer Disease
MeSH Terms: conditions — Aphasia, Primary Progressive; Anomia; Alzheimer Disease

ARMS (2):
- Phonological, Orthographic, Untrained (Experimental)
  Interventions: Behavioral: Phonological; Behavioral: Orthographic; Behavioral: Untrained
- Semantic, Lexical, Untrained (Experimental)
  Interventions: Behavioral: Semantic; Behavioral: Lexical; Behavioral: Untrained

INTERVENTIONS:
Behavioral: Phonological — This treatment involves picture viewing and word repetition.
  Arms: Phonological, Orthographic, Untrained
Behavioral: Orthographic — This treatment involves picture viewing, reading, and writing.
  Arms: Phonological, Orthographic, Untrained
Behavioral: Semantic — This treatment involves learning about the semantic features (meaning) of each trained word.
  Arms: Semantic, Lexical, Untrained
Behavioral: Lexical — This treatment involves learning about the lexical features (letters and sounds) of each trained word.
  Arms: Semantic, Lexical, Untrained
Behavioral: Untrained — These words are not trained during the treatment phase.

SUMMARY:
The goal of this study is to remediate word-finding problems in patients who have Primary Progressive Aphasia (PPA) or Alzheimer's Disease and to delay the further progression of word-finding impairment. The current approach is novel in that it contains a prophylaxis component in which the investigators attempt to strengthen neural connections that remain functional, making them more resistant to degradation as the disease progresses. While the study is specific in its targeting of word-finding problems, a successful outcome would bode well for other studies aimed at prevention or reversal of declining cognitive functions in dementia. One set of participants with PPA will receive practice with picture naming in two conditions: viewing the picture and repeating the name; and viewing the picture with its written name, plus reading and writing the name. Another set of participants with PPA or Alzheimer's Disease will be trained in two different conditions: learning about the word's semantic features (meaning); and learning about the word's lexical features (letters and sounds). Naming of pictures trained in each of these conditions will be compared, at three time intervals post-training, with naming of pictures tested before the study but never trained. It is predicted that the pairing of the picture with its written name, combined with the motor task of writing the name, will result in a greater ability to name the picture at a later date than simple practice viewing the picture and repeating the name. Furthermore, it is predicted that participants who have difficulty understanding concepts will be more likely to respond to semantic treatment, while participants who have difficulty connecting words with concepts will be more likely to respond to lexical treatment.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Primary Progressive Aphasia (PPA; including Frontotemporal Dementia, Semantic Dementia, or a similar condition) or Diagnosis of Alzheimer's Disease
* At least 10 years of education
* Ability to follow spoken instructions
* Medically stable
* First language is English, or fluent in English since childhood
* Willing to participate over a period of two years

Exclusion Criteria:

* No history of additional neurological problems
* No history of substance abuse or psychiatric problems

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2011-11 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Change in picture naming accuracy for words within each treatment condition during treatment | baseline, 7 months
  The change in picture naming accuracy for trained words will be compared with the change in picture naming accuracy for words that were tested at baseline but never trained during the treatment phase.

SECONDARY OUTCOMES:
Change in picture naming accuracy for words within each treatment condition between baseline and first follow-up assessment | baseline, 14 months
  The change in picture naming accuracy for trained words will be compared with the change in picture naming accuracy for words that were tested at baseline but never trained during the treatment phase.
Change in picture naming accuracy for words within each treatment condition between baseline and second follow-up assessment | baseline, 21 months
  The change in picture naming accuracy for trained words will be compared with the change in picture naming accuracy for words that were tested at baseline but never trained during the treatment phase.

CONTACTS AND LOCATIONS:
Overall Officials: Aaron Meyer, PhD, Principal Investigator — Georgetown University
Locations (2):
- United States (2):
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - Johns Hopkins University, Baltimore, Maryland

REFERENCES:
- [Derived] Suh S, Friedman RB, Meyer AM, Snider SF, Sebastian R, Tippett DC. Picture Description and Functional Communication Rating Correlates in Variants of Primary Progressive Aphasia. Aphasiology. 2025 May 28:10.1080/02687038.2025.2510327. doi: 10.1080/02687038.2025.2510327. Online ahead of print. PMID 40857539
- See also: Center for Aphasia Research and Rehabilitation website — http://faculty.georgetown.edu/friedmar/carr.html